CLINICAL TRIAL: NCT06964295
Title: Comparison of First Attempt Success in Nasotracheal Intubation Using Macintosh Videolaryngoscope vs. Flexible Bronchoscope: a Randomized Controlled Trial
Brief Title: Comparison of First Attempt Success in Nasotracheal Intubation Using Macintosh Videolaryngoscope vs. Flexible Bronchoscope
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2503-041-1621
Record Dates: First submitted 2025-04-23; First posted 2025-05-09 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-04

CONDITIONS: Intubation Complication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Videolaryngoscope Group (Experimental)
  Interventions: Device: Macintosh videolaryngoscope
- Flexible Bronchoscope Group (Active Comparator)
  Interventions: Device: Flexible bronchoscope

INTERVENTIONS:
Device: Macintosh videolaryngoscope — Used to perform nasotracheal intubation under general anesthesia. The Macintosh videolaryngoscope is introduced orally to visualize the glottis, and a preformed nasotracheal tube is inserted through the nostril.
  Arms: Videolaryngoscope Group
Device: Flexible bronchoscope — Used to perform nasotracheal intubation under general anesthesia. The bronchoscope is inserted through a lubricated nasotracheal tube and advanced into the trachea.
  Arms: Flexible Bronchoscope Group

SUMMARY:
Participants are randomly assigned to two groups: one group undergoes nasotracheal intubation using a videolaryngoscope, while the other group undergoes nasotracheal intubation using a flexible bronchoscope. The primary outcome is the first-attempt success rate, assessed at the time of tracheal tube placement. Additional outcomes include the degree of subglottic injury upon extubation, and the incidence and severity of sore throat and hoarseness at 1 hour and 24 hours postoperatively, as well as overall intubation success rates.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years or older
* Undergoing ear, nose, and throat (ENT) surgery requiring nasotracheal intubation

Exclusion Criteria:

* Refusal to participate in the study
* History of gastroesophageal reflux disease
* History of surgery or radiation therapy involving the upper airway
* Presence of severely loose teeth

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2026-05-07 (Estimated); Study Completion 2026-05-07 (Estimated)

PRIMARY OUTCOMES:
First-attempt success rate of nasotracheal intubation | At the time of tracheal intubation
  The proportion of patients in whom nasotracheal intubation is successfully completed on the first attempt, comparing the videolaryngoscope group with the flexible bronchoscope group.

SECONDARY OUTCOMES:
Degree of subglottic injury | At the time of extubation
  Graded from 0 to 3 using a flexible bronchoscope. Higher scores mean a worse outcome (more severe subglottic injury).
Postoperative sore throat severity | 1 hour and 24 hours postoperatively
  Assessed using the Numeric Rating Scale (0-10) at 1 and 24 hours after surgery.
Incidence of postoperative hoarseness | 1 hour and 24 hours postoperatively
  Presence or absence of hoarseness evaluated at 1 hour and 24 hours postoperatively.
Cormack-Lehane grade | At the time of tracheal intubation
  Grading recorded during intubation to evaluate glottic exposure.
Changes in blood pressure | Within 5 minutes before and after intubation
  Changes in blood pressure recorded before and after tracheal intubation.
POGO score | At the time of tracheal intubation
  Visualization scores recorded during intubation to evaluate glottic exposure. The score ranges from 0% (no glottic visualization) to 100% (full view of the glottis). Higher scores indicate a better outcome (better visualization).
Changes in heart rate | Within 5 minutes before and after intubation
  Changes in heart rate recorded before and after tracheal intubation.
Changes in saturation | Within 5 minutes before and after intubation
  Changes in SpO₂ recorded before and after tracheal intubation.
Changes in bispectral value | Within 5 minutes before and after intubation
  Changes in BIS values recorded before and after tracheal intubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea